CLINICAL TRIAL: NCT03213288
Title: The Effects of Bilberry Fruit and Black Rice Derived Anthocyanins on Lipid Status in Adults
Brief Title: Bilberry Fruit and Black Rice Derived Anthocyanins on Lipid Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quadram Institute Bioscience (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: IFR01/2017
Record Dates: First submitted 2017-07-05; First posted 2017-07-11 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Delphinidin type anthocyanins (Active Comparator): Bilberry extract
  Interventions: Dietary Supplement: Delphinidin type anthocyanins
- Cyanidin type anthocyanins (Active Comparator): Black rice extract
  Interventions: Dietary Supplement: Cyanidin type anthocyanins
- Placebo (Placebo Comparator): No anthocyanins
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Delphinidin type anthocyanins — Bilberry extract containing Delphinidin type anthocyanins
  Arms: Delphinidin type anthocyanins
Dietary Supplement: Cyanidin type anthocyanins — Black rice extract containing Cyanidin type anthocyanins
  Arms: Cyanidin type anthocyanins
Dietary Supplement: Placebo — No anthocyanins
  Arms: Placebo

SUMMARY:
The primary aim of this study is to directly compare the two major types of anthocyanins found in the diet (cyanidin-type and delphinidin-type) on lipid status in adults.

DETAILED DESCRIPTION:
Human intervention trials with anthocyanin-rich berry fruits/extracts such as whole strawberries, elderberry juice and whortleberry extracts, and purified anthocyanins from a mixture of blackcurrant and bilberry have been shown to beneficially alter biological markers for CVD risk, with beneficial effects on lipid profiles common across these studies.

In a randomized 3 phase crossover study we aim to recruit 50 participants (men and women) aged 45 years or more with a higher than optimal blood cholesterol level to consume capsules containing (i) 320 mg anthocyanins derived from bilberry fruit (delphinidin type), (ii) 320 mg anthocyanins derived from black rice (cyanidin type) and (iii) a placebo control. Each treatment will be ingested for 28 days with a wash-out period of 4 weeks in-between. Blood samples will be collected at the start and end of each 28-day treatment period to assess lipid status. In a subset of participants we will also investigate the relationship between bilberry and black rice anthocyanin ingestion on RNA expression profiles that are known to be involved in atherosclerosis, non-alcoholic fatty liver disease and reverse cholesterol transport as well as faecal excretion of bile acids and lipids.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 45 years of age
* Total cholesterol ≥ 5.0 mmol/L

Exclusion Criteria:

* Smokers (or stopped smoking for less than 3 months)
* Medical conditions that are judged to affect the primary outcome measure for this study or which may compromise the well-being of the participant e.g. diabetes.
* Prescribed and non-prescribed medications that may affect the primary outcome measure for this study e.g. lipid lowering therapy
* Dietary supplements judged to affect the study data unless the participant is willing to discontinue them for 4 weeks preceding the start of the study and for the duration of the study
* Use foods for lowering cholesterol e.g. benecol, flora proactive
* Regular/recent use of colonic irrigation or other bowel cleansing techniques.
* Intend to change the normal use of pre or probiotics during the study (only applies to those collecting faecal samples)
* Bowel movements ≤ 3 times per week (only applies to those collecting faecal samples)
* Gastro-intestinal diseases (excluding hiatus hernia unless symptomatic or study intervention/procedure is contra-indicated).
* Parallel participation in another research project which involves dietary intervention
* Participation in another research project which has involved blood sampling within the last four months unless the total amount of combined blood from both studies does not exceed 470 ml.
* Has donated or intends to donate blood within 16 weeks prior to or during the study period.
* Any person related to or living with any member of the study team
* Lack of capacity to provide written informed consent
* Are pregnant or have been pregnant within the last 12 months

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
LDL cholesterol | 28 days
  Serum lipid status

SECONDARY OUTCOMES:
Total/HDL cholesterol and triglycerides | 28 days
  Serum lipid status and faecal excretion of lipids
Cholesterol efflux capacity | 28 days
  Cholesterol metabolism
PON-1 activity | 28 days
  Cholesterol metabolism
Bile acids and derivatives | 28 days
  Plasma bile acid status and faecal excretion of bile acids
Glucose, fructosamine and insulin | 28 days
  glycaemic control
MicroRNA expression | 28 days
  MicroRNA's implicated in atherosclerosis, non-alcoholic fatty liver disease and reverse cholesterol transport

CONTACTS AND LOCATIONS:
Overall Officials: Paul Kroon, Principal Investigator — Quadram Institute Bioscience
Locations (1):
- Quadram Institute Bioscience, Norwich, United Kingdom

IPD SHARING:
Plan to Share IPD: No